CLINICAL TRIAL: NCT00218985
Title: Exercise-training Before Coronary Artery Bypass Graft (CABG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TRIM 158-04
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Angina; Coronary Artery Disease
Keywords: Aerobic capacity; Exercise training; CABG; Endothelial function
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise training (Experimental)
  Interventions: Behavioral: Exercise training
- physician's advice (No Intervention): patients follow their physician's advice in regard to physical activity.

INTERVENTIONS:
Behavioral: Exercise training — Intensity controlled exercise training before the scheduled bypass surgery
  Arms: exercise training

SUMMARY:
The aim is to evaluate the effect of exercise training upon endothelial function in the mammary artery of patients who are scheduled for CABG, as well as study the functional properties of single cells isolated from a small biopsy of the left ventricle obtained during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for CABG both with and without heart failure

Exclusion Criteria:

* Unstable angina
* Unable to walk on a treadmill (except those with heart failure who only will serve as a reference group)
* Participation in another study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular function and quality of life | Before and up to 1 year after intervention

SECONDARY OUTCOMES:
Structure and function of cardiomyocytes | After the intervention period
Cardiomyocyte structure and function | after the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisloff, Ph.D, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Smenes BT, Baekkerud FH, Slagsvold KH, Hassel E, Wohlwend M, Pinho M, Hoydal M, Wisloff U, Rognmo O, Wahba A. Acute exercise is not cardioprotective and may induce apoptotic signalling in heart surgery: a randomized controlled trial. Interact Cardiovasc Thorac Surg. 2018 Jul 1;27(1):95-101. doi: 10.1093/icvts/ivx439. PMID 29447379